CLINICAL TRIAL: NCT03493750
Title: Oral Evaluation by the Nurses From the Office of Access to Healthcare ("PASS") for Vulnerable People as a Vector for the Detection of Oral Diseases to Improve Access to the Appropriate Healthcare Branch - PASSDENT Study
Brief Title: Oral Evaluation by the Nurses From the Office of Access to Healthcare ("PASS") for Vulnerable People - PASSDENT Study
Acronym: PASSDENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P_2015_003; 2015-A01878-41 (Other: ANSM (French National Drug Safety Agency))
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Homeless and Low Incomes People, Refugees

STUDY DESIGN:
Intervention Model Description: Impact of an oral evaluation realized by a nurse combined with a questionnaire (the healthplan guide)
Who Masked: Care Provider
Masking Description: Dentists are masked of the patient group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthplan guide alone (No Intervention): Nurse applies the daily-practice questionnaire called "Healthplan guide" to screen and identify people with dental diseases, among those in vulnerable situation, and to sensitize them about the importance of oral hygiene and how to improve it.
  After that, the nurse has to state if, from her/his point of view the patient needs dental care or not. Whatever the answer, the nurse makes an appointment to a dental practice, in the 30 following days, and gives it to the patient with a free bus ticket. Randomization is done at that time.
  The dentist, blinded of the patient's group, makes a dental exam and says if the patient needs dental care or not.
  If care are indicated, they will be organized but outside this trial.
- Oral and dental evaluation (Experimental): After application of the "Healthplan guide", nurse statement of the need of dental care or not, making of an appointment to the dental practice and gift of a free bus ticket, if the patient is randomized in the experimental group, the nurse completes the evaluation with a mouth inspection in order to count missing, coloured, injured teeth, and evaluate dental plaque, halitosis, inflammatory gums, mucosal injuries, low masticatory surface. At the end of this exam, the nurse has to state again if, from her/his point of view the patient needs dental care or not.
  The dentist, blinded of the patient's group, makes a dental exam and says if the patient needs dental care or not.
  If care are indicated, they will be organised but outside this trial.
  Interventions: Other: Oral and dental evaluation

INTERVENTIONS:
Other: Oral and dental evaluation — Mouth inspection done by a nurse, in order to count missing, coloured, injured teeth, and evaluate dental plaque, halitosis, inflammatory gums, mucosal injuries, low masticatory surface.
  Arms: Oral and dental evaluation

SUMMARY:
Oral health is defined as the state of being free from dental or periodontal diseases and discomfort of oral cavity. WHO considers that oral hygiene is a major public health problem whatever the countries (developed, developing, and underdeveloped).

The two main local medical problems are dental caries and periodontal diseases. Without appropriate treatments, both diseases can lead to local functional and esthetic damages, and can also have some negative repercussions on health.

Studies showed that there are great social disparities among people concerned by oral health issues. People in vulnerable situations (homeless and low incomes people, refugees) had less recourse to dental care. Those who consult do it less often and later. Reasons are mainly cost related, but also people in vulnerable situation don't perceive dental care as an important matter and don't know where and how to ask for help for having dental care.

PASS (french acronym for "Office of Access to Healthcare") departments, setting in both private and public health institutions, are intended to facilitate the access to care and the support of people in vulnerable situations, and their accompaniment in the steps necessary for the recognition of their rights.

Nurses of the Annecy PASS department had developed a questionnaire called "healthplan guide" that aim at helping them to screen and identify people with dental diseases among those in vulnerable situation, and to sensitize them about the importance of oral hygiene and how to improve it. This questionnaire is use in daily practice.

This study hypothesizes that more patients will be sensitized to benefit a dental examination in a dental practice if nurses use the "healthplan guide" questionnaire combined with an oral and dental evaluation.

DETAILED DESCRIPTION:
Oral health is defined as the state of being free from dental or periodontal diseases and discomfort of oral cavity. WHO considers that oral hygiene is a major public health problem, as regard to number of people involved and the consequences either local (pain, functional deteriorations, teeth loss) or general (decreased quality of life, lower health status and increased mortality rate).

The two main local medical problems are dental caries and periodontal diseases ; among adults this is a major public health problem whatever the countries. Furthermore, the cost of these diseases is high, for example ranking fourth in developed countries health costs.

Dental caries is the most prevalent disease worldwide. The local production of organics acids by cariogenic bacteria located in the dental plaque, leading to the reduction of local pH, is responsible for enamel demineralisation and tooth decay. The local production of organic acids is due to the metabolism of fermentable sugars by bacteria of the dental plaque, saccharose being considered as the most cariogenic one. Dental caries occur when pH modification is durable. First, tooth decay affects only enamel and can be cured if appropriate measures favorising remineralisation are used. Second, when the enamel is totally destroyed, the hole inside dentin is irreversible and requires specific care.

Periodontal disease is also due to bacterias located in the dental plaque, with first, a local inflammatory reaction in the soft tissues of the tooth (gum and alveolar bone) that, second, lead to their destruction. This is a long lasting course disease.

Without appropriate treatments, both diseases can lead to local functional and esthetic damages, and can also have some negative repercussions on health, putting the patient at a higher risk of infectious endocarditis, cardiovascular or bronchopulmonary diseases, preterm deliveries, pre-eclampsias, poor control of diabetes, or increased rheumatoid arthritis exacerbations.

Furthermore, some other diseases are likely to favor bucco-dental diseases, such as diabetes, or immunosuppressive diseases for example AIDS.

Some medicines, particularly those inducing xerostomia increase the development of bucco-dental diseases. Alcohol and tobacco consumption is known to be an important risk factor.

Studies showed that there are great social disparities among people concerned by oral health issue. For example, people with low incomes have more missing teeth, dental caries needing care or avulsions, parodontal diseases and deficient oral hygiene. People in vulnerable situations (homeless and low incomes people, refugees) have less recourse to dental care. Those who consult do it less often and later. Reasons are mainly cost related, but also people in vulnerable situation don't perceive dental care as an important matter in absence of pain and don't know where and how to ask for help for having dental care.

In France, in 1998 an act (Loi d'orientation du 29 juillet 1998 "relative à la lutte contre les exclusions") implemented the permanent access to health care for people in vulnerable situations and created departments called PASS (french acronym for "Office of Access to Healthcare"). These structures, setting in both private and public health institutions, are intended to facilitate the access to care of people in vulnerable situations, and to support them throughout all the steps required to obtain recognition of their rights.

PASS-Annecy department was created in 2003 in Annecy hospital. In 2010, the French High Authority for Public Health published some recommendations on caries prevention; development of dental consultations for people in vulnerable situation in local structures such as PASS were encouraged.

After severe infections (endocarditis and face cellulitis) in two homeless people in Annecy hospital, nurses of the Annecy PASS department had developed a questionnaire called "healthplan guide" that aim at helping them to screen and identify people with dental diseases among those in vulnerable situation, and to sensitize them about the importance of oral hygiene and how to improve it. This questionnaire is use in daily practice. Nevertheless, despite sensitization with the "healthplan guide" use, few people among vulnerable one's went to the dental practice after the nurses made them an appointment.

This study hypothesizes that more patients will be sensitized to have a dental examination in dental practice if nurses will do an oral and dental evaluation combined with the use of the "healthplan guide" questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* people helped by the PASS department
* seen for the first or the second time in the PASS department
* older than 18 years old
* able to read and understand one of the following languages: French, English or the Albanian language of Kosovo
* with or without insurance coverage
* who had given their informed consent

Exclusion Criteria:

* people without any identity document
* psychiatric disease compromising the comprehension of the study
* edentulous people or those with whole dental prosthesises
* people who intend to leave the Annecy area within few days
* people requiring emergency care whatever the reason
* people not able to go alone to the dental practice
* pregnant or lactating women
* people with law protection (i.e. under legal guardianship or curators)
* people suffering from violence injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Impact of an oral evaluation realized by a nurse combined with a questionnaire compared with the use of the questionnaire alone | 60 days
  Rate of people who go to the dental practice after an appointment booked by the nurse of the PASS structure

SECONDARY OUTCOMES:
Oral health care status of the study population | 1 day
  Oral evaluation and oral hygien index done by dentists with only one evaluation form
Relevance of the nurse in identifying patients requiring oral care | 1 day
  Comparison of nurse and dentist evaluations concerning the need of dental care
Quality of the oral evaluation done by trained nurses, in the experimental group only | 1 day
  Agreement between nurse and dentist concerning number and location of missing, coloured, injured teeth (according to the World Dental Federation two-digit notation), dental plaque, halitosis, inflammatory gums, mucosal injuries, low masticatory surface.

CONTACTS AND LOCATIONS:
Overall Officials: Louisa Chevaleyre, Nurse, Principal Investigator — CH Annecy Genevois
Locations (7):
- France (7):
  - ADOMA, Annecy
  - Centre d'hébergement et de réinsertion sociale Saint-François, Annecy
  - L'Herminette, Annecy
  - L'Intervalle, Annecy
  - La Halte, Annecy
  - Ma Bohème, Annecy
  - CH Annecy Genevois, Pringy

IPD SHARING:
Plan to Share IPD: No